CLINICAL TRIAL: NCT05380661
Title: Heart Rate Variability During Urinary Bladder Catheterization in Individuals With Spinal Cord Injury: Anxiety Versus Sensory Discomfort
Brief Title: Heart Rate Variability and Anxiety During Urinary Bladder Catheterization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: ConvaTec Inc. (Industry); Vancouver Coastal Health (Other Government); International Collaboration on Repair Discoveries (Other)
Responsible Party: Principal Investigator, Andrei Krassioukov, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: H22-00971
Record Dates: First submitted 2022-05-05; First posted 2022-05-19 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Spinal Cord Injuries; Urinary Bladder, Neurogenic; Anxiety State; Catheter Complications; Autonomic Dysreflexia
Keywords: Intermittent Catheterization
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic; Anxiety Disorders; Autonomic Dysreflexia | interventions — Intermittent Urethral Catheterization

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants blinded to order of catheterization procedures conducted by the urology nurse.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individuals with motor-complete SCI (Experimental): Individuals with motor sensory complete injury (AIS A/B)
  Interventions: Procedure: Self-catheterization; Procedure: Catheterization performed by urology nurse, participant blinded to time of procedure; Procedure: Catheterization performed by urology nurse, participant aware of time of procedure
- Individuals with motor-incomplete SCI (Experimental): Individuals with motor sensory incomplete injury (AIS C/D)
  Interventions: Procedure: Self-catheterization; Procedure: Catheterization performed by urology nurse, participant blinded to time of procedure; Procedure: Catheterization performed by urology nurse, participant aware of time of procedure

INTERVENTIONS:
Procedure: Self-catheterization — Participants will perform self-catheterization, following the same routine for intermittent catheterization at home
Procedure: Catheterization performed by urology nurse, participant blinded to time of procedure — Participant will undergo procedure to completely empty bladder; Participant in supine position, and resting blood pressure and heart rate will be recorded for period of 5 minutes prior to catheterization; Perineum and genital areas will be draped and they will be not aware about exact timing of catheterization Catheterization will be conducted following standard clinic procedure by experience urology nurse.
Procedure: Catheterization performed by urology nurse, participant aware of time of procedure — Participant will undergo procedure to completely empty bladder; Participant in supine position, and resting BP and HR will be recorded for period of 5 minutes prior to catheterization; Perineum and genital areas will be visible to participant and they will be fully aware about exact timing of catheterization Catheterization will be conducted following standard clinic procedure by experience urology nurse.

SUMMARY:
This is a prospective, randomised study investigating the physical and psychological experience of intermittent catheterization in adult individuals following spinal cord injury (SCI).

DETAILED DESCRIPTION:
Given that intermittent catheterization is the recommended method of bladder management in individuals with SCI, it is crucial that the potentially negative cardiovascular and psychological responses to this procedure are examined. Individuals will undergo self-catheterization, then two standard of care catheterization procedures performed by an experienced urology nurse, while either blinded to or aware of time of catheterization. Continuous cardiovascular monitoring will be in place throughout all three procedures. Assessment of anxiety will be administered pre- and post- each procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-70 years of age
* Any chronic traumatic SCI with either motor sensory complete injury (AIS A/B, N=10) or motor sensory incomplete injury (AIS B/D, N=10).
* At least 1 year post injury, and at least 6 months from any spinal surgery
* Hand function sufficient to perform intermittent catheterization for management of urinary bladder drainage
* Must provide informed consent and be able to understand and complete study-related questionnaires (must be able to understand and speak English or have access to an appropriate interpreter as judged by the investigator)
* Willing and able to comply with clinic visit and study-related procedures

Exclusion Criteria:

* Signs or known current urinary tract infection, or other inflammatory conditions of bladder/urethra
* Currently taking beta blockers or other medications that may affect heart rate
* History of ureteral injury
* History of any urinary diversion procedures, including but not limited to bladder augmentation, cystectomy, neo bladder, pouch reservoir, ileal conduit, Mitrofanoff appendicovesicostomy
* For women of childbearing potential, currently pregnant
* A member of the investigational team or his/her immediate family Presence of severe acute medical issue and use of any specific medication or treatment that, in the investigator's judgement, would adversely affect the participant's participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure (BP) during self-catheterization | During self-catheterization
  Systolic and diastolic BP (mmHg) will be measured continuously (beat-by-beat) via finger photoplethysmography, corrected to brachial pressure. BP will be measured 5 minutes prior to and then throughout the self-catheterization procedure.
Heart rate (HR) during self-catheterization | During self-catheterization
  HR (BPM) will be recorded continuously via one-lead electrocardiogram. HR will be measured 5 minutes prior to and then throughout the self-catheterization procedure.
BP during catheterization performed by urology nurse, participant blinded to time of procedure | During catheterization performed by urology nurse, participant blinded to time of procedure
  Systolic and diastolic BP (mmHg) will be measured 5 minutes prior to and then throughout the standard of care catheterization performed by an experienced urology nurse, while the participant is blinded to time of procedure.
HR during catheterization performed by urology nurse, participant blinded to time of procedure | During catheterization performed by urology nurse, participant blinded to time of procedure
  HR (BPM) will be measured 5 minutes prior to and then throughout the standard of care catheterization performed by an experienced urology nurse, while the participant is blinded to time of procedure.
BP during catheterization performed by urology nurse, participant aware of time of procedure | During catheterization performed by urology nurse, participant aware of time of procedure
  Systolic and diastolic BP (mmHg) will be measured 5 minutes prior to and then throughout the standard of care catheterization performed by an experienced urology nurse, while the participant is aware of time of procedure.
HR during catheterization performed by urology nurse, participant aware of time of procedure | During catheterization performed by urology nurse, participant aware of time of procedure
  HR (BPM) will be measured 5 minutes prior to and then throughout the standard of care catheterization performed by an experienced urology nurse, while the participant is aware of time of procedure.
Change in state anxiety in the context of self-catheterization (STAIS-5) | 5 minutes before and 5 minutes after self-catheterization
  The State-Trait Anxiety Inventory - State, 5 item version (STAIS-5) will be used to measure participants' state anxiety prior to and after self-catheterization. Sum score of the STAIS-5 will be calculated, which ranges between 5 to 20, with higher score indicating greater state anxiety.
Change in state anxiety in the context of catheterization performed by urology nurse, participant blinded to time of procedure (STAIS-5) | 5 minutes before and 5 minutes after catheterization performed by urology nurse, participant blinded to time of procedure
  The STAIS-5 will be used to measure participants' state anxiety prior to and after catheterization procedure performed by an experienced urology nurse, while the participant is blinded to time of procedure. Sum score of the STAIS-5 will be calculated, which ranges between 5 to 20, with higher score indicating greater state anxiety.
Change in state anxiety in the context of catheterization performed by urology nurse, participant aware of time of procedure (STAIS-5) | 5 minutes before and 5 minutes after catheterization performed by urology nurse, participant aware of time of procedure
  The STAIS-5 will be used to measure participants' state anxiety prior to and after catheterization procedure performed by an experienced urology nurse, while the participant is aware of time of procedure. Sum score of the STAIS-5 will be calculated, which ranges between 5 to 20, with higher score indicating greater state anxiety.

SECONDARY OUTCOMES:
Baseline trait anxiety | During screening
  The 7-item General Anxiety Disorder (GAD) scale will be used to measure participants' anxiety. The GAD-7 sum score will be calculated, ranging from 0 to 21, with higher score indicating more severe anxiety symptoms.
Change in state anxiety in the context of self-catheterization (GA-VAS) | 5 minutes before and 5 minutes after self-catheterization
  The Global Anxiety-Visual Analogue Scale (GA-VAS) will be used to measure participants' state anxiety prior to and after self-catheterization. Rating can range between 0 to 10, with higher rating on the GA-VAS indicates greater state anxiety.
Change in state anxiety in the context of catheterization performed by urology nurse, participant blinded to time of procedure (GA-VAS) | 5 minutes before and 5 minutes after catheterization performed by urology nurse, participant blinded to time of procedure
  The GA-VAS will be used to measure participants' state anxiety prior to and after catheterization procedure performed by an experienced urology nurse, while the participant is blinded to time of procedure. Rating can range between 0 to 10, higher rating on the GA-VAS indicates greater state anxiety.
Change in state anxiety in the context of catheterization performed by urology nurse, participant aware of time of procedure (GA-VAS) | 5 minutes before and 5 minutes after catheterization performed by urology nurse, participant aware of time of procedure
  The GA-VAS will be used to measure participants' state anxiety prior to and after catheterization procedure performed by an experienced urology nurse, while the participant is aware of time of procedure. Higher rating on the GA-VAS indicates greater state anxiety.
Change in heart rate variability (HRV) during self-catheterization | During self-catheterization
  HRV will be calculated from continuous ECG recording
Change in heart rate variability (HRV) during catheterization performed by urology nurse, participant blinded to time of procedure | During catheterization performed by urology nurse, participant blinded to time of procedure
  HRV will be calculated from continuous ECG recording
Change in heart rate variability (HRV) during catheterization performed by urology nurse, participant aware of time of procedure | During catheterization performed by urology nurse, participant aware of time of procedure
  HRV will be calculated from continuous ECG recording

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Krassioukov, MD,PhD,FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- Blusson Spinal Cord Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided